CLINICAL TRIAL: NCT04821661
Title: Duration of Bloodstream Infection as Measured by Conventional Cultures Compared With Novel Culture Independent Systems and Persistence of Biomarkers Associated With Severe Infection
Brief Title: T2 and SeptiCyte RAPID Duration Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Metro North Hospital and Health Service (Unknown); Pathology Queensland (Unknown)
Responsible Party: Principal Investigator, Professor David L. Paterson, Professor, The University of Queensland
Other Study IDs: HREC/2021/QRBW/70126
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Bacteremia
Keywords: Bacteraemia; Gram-negative Bacteremia; Bacterial Infections; T2 magnetic resonance assay; SeptiCyte RAPID
MeSH Terms: conditions — Bacteremia; Toxemia; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infection with bacteria and other germs in the blood can be deadly. How long germs stay in the blood is important for two reasons. The first is that if they stay in the blood for many days it is a sign that antibiotics may need to be changed. The second is that if they stay in the blood for only a short time it may give doctors confidence to switch to tablets and consider early discharge from hospital. This study is evaluating the diagnostic and prognostic performance of two novel technologies when used to measure the duration of the bloodstream infection.

DETAILED DESCRIPTION:
Bloodstream infection is highly significant and is associated with mortality rates of between 10 and 25%.

For some infection types (for example, Staphylococcus aureus) a longer duration of bacteria being present in the blood is linked to higher mortality. With traditional microbiologic techniques, bloodstream infection with gram-negative bacteria is usually quite brief. However, new culture independent bacteraemia detection systems (such as T2 magnetic resonance assay) are more sensitive than traditional blood culture systems and may show that gram-negative bacteraemia is more prolonged in some patients than has previously been thought. This observational study will investigate the correlation between the duration of bloodstream infection by mean of traditional blood culture techniques with:

1. Duration of the bloodstream infection by mean of the T2 magnetic resonance assay, a new culture independent bacteraemia detection system.
2. Persistence of inflammation as measured by the SeptiCyte RAPID test, a host response assay able to differentiate infectious from sterile inflammation.

The study will also correlate each measure of the duration of bacteraemia with microbiological and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have proven bloodstream infection with any T2-on panel pathogen (Enterococcus faecium, S. aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa, Escherichia coli and Candida spp.)

Exclusion Criteria:

* Palliative care approach
* Failure to give written informed consent (by patient or their legal representative)
* Polymicrobial index blood culture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Royal Brisbane and Women's Hospital, Caboolture Hospital and Redcliffe Hospital who have bacteria or yeast in the blood identified by the MALDI-TOF MS and Gram stain respectively
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Duration of bloodstream infection measured by conventional blood cultures and the T2 magnetic resonance assay | Days 1-4
  The T2 system is a new diagnostic detection method utilizing miniaturized magnetic resonance technology. The T2 system has been shown to quickly and accurately identify molecular targets within patient samples without the need for purification or extraction of target molecules from the sample. It does not require bacterial culture and can detect organisms as low as 1 CFU/mL in whole blood. The study will compare the duration of detectable pathogens in the bloodstream as measured by the T2 with the duration of bloodstream infection according to conventional cultures
Persistent infection defined as metastatic infection and lack of source control | Days 1-4
  The study will explore the correlation between the duration of detectable pathogens in the bloodstream as measured by the T2 (duration of T2emia) and the presence of persistent infection

SECONDARY OUTCOMES:
Short-term clinical outcome (SOFA success) | Days 1-7
  The study will explore the correlation between the duration of detectable pathogens in the bloodstream as measured by the T2 (duration of T2emia) and short-term clinical outcome. A "successful short-term outcome" or "SOFA success" is defined as survival for the first 7 days from BSI onset with a stable or decreased Sequential Organ Failure Assessment (SOFA) score (for ICU patients) or modified SOFA score (for non-ICU patients), defined as follows: if the baseline SOFA/mSOFA >=3, a decrease of at least 30% in that score, if the baseline SOFA/mSOFA <3, a stable or decreased SOFA/mSOFA score. Patients discharged before day 7 will be assumed to have improved SOFA scores. The lack of "SOFA success" will be defined "SOFA failure".
Long-term clinical outcome | 6-months from the index BSI
  The study will explore the correlation between the duration of detectable pathogens in the bloodstream as measured by the T2 (duration of T2emia) and long-term clinical outcomes. A "successful long-term outcome" is defined as survival for the first 6 months from the BSI onset and maintenance of the baseline functional performance status defined by the functional bloodstream infection score (FBIS) score 7 days prior to the BSI onset.
Persistent infection | Day 1-4
  SeptiCyte is a host-response assay able to differentiate infectious from sterile inflammation by providing a score (SeptiScore) from 1-15. It is approved for the diagnosis of sepsis in ICU patients. Whether SeptiScore may have a role in diagnosing the persistence of the infection in patients with proven BSI is unknown. The study will explore the performance of SeptiScore in diagnosing persistent infection including persistent BSI and metastatic infection

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Caboolture Hospital, Brisbane, Queensland
  - Redcliffe Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland